CLINICAL TRIAL: NCT01306812
Title: Risk Factors for Alcohol Abuse and Deviant Behaviour - Biochemical and Molecular Studies in Adolescents From Swedish County
Brief Title: Survey of Adolescent Living in Vestmanland
Acronym: SALVe
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Jerzy Leppert, Medical Faculty , Uppsala universitet
Other Study IDs: SALVe
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-03

CONDITIONS: Alcohol Abuse; Criminalism; Depression
Keywords: Adolescent; Alcohol; Criminology; Genes; Environment; Mono amine Oxidase; Serotonin; Social Support
MeSH Terms: conditions — Alcoholism; Depression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The interaction of MAO-A genotype and psychosocial risk, in relation to male adolescent criminality The interaction of 5-HTTLPR genotype and psychosocial risk in relation to excessive adolescent alcohol consumption The interaction of 5-HTTLPR genotype and psychosocial risk in relation to depressive symptoms among adolescents The interaction of MAO-A genotype and psychosocial risk, in relation to female adolescent criminality

ELIGIBILITY:
Inclusion Criteria:

All students present in school class during survey

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 16 and 19-year-olds school students in county of Vestmanland.
Sampling Method: Probability Sample
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Västerås, Vasteras, Sweden